CLINICAL TRIAL: NCT02676128
Title: Mobile Health Application to Improve HIV Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH108431 (NIH)
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: HIV; Medication Adherence; Mobile Health
Keywords: HIV; Medication Adherence; Mobile Health
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile Health ART Adherence Application (mARTAA) (Experimental): mARTAA will use a smartphone-delivered application developed by Twine Health, Inc.
  Interventions: Behavioral: Twine Collaborative Care Application
- Face-to-Face ART Adherence Intervention (Active Comparator): A single face-to-face ART adherence intervention will be administered.
  Interventions: Behavioral: Information-Motivation-Behavioral Skills Model of ART Adherence

INTERVENTIONS:
Behavioral: Twine Collaborative Care Application — This application features a 24-hour medication clock that displays ART dosing schedule and allows participants to record the doses taken. It also features an interactive health coaching feature which will be used to provide support, encouragement, and resources to participants.
  Arms: Mobile Health ART Adherence Application (mARTAA)
Behavioral: Information-Motivation-Behavioral Skills Model of ART Adherence — Combines brief motivational interviewing, cognitive behavior therapy, and problem-solving skills to help participants formulate and follow ART adherence goals.
  Arms: Face-to-Face ART Adherence Intervention

SUMMARY:
Inadequate adherence to antiretroviral therapy (ART) can impede successful viral suppression and consequently lead to negative health consequences. This study aims to refine and test the efficacy of a mobile health ART adherence application (ARTAA), delivered over a smartphone, with helping individuals improve their ART adherence.

DETAILED DESCRIPTION:
The CDC estimates that 1.1 million people living in the U.S. are infected with HIV [1]. Only a quarter of person living with HIV (PLWH) successfully keep the virus under control [2]. Medication non-adherence is a significant contributor to unsuccessful viral suppression; a recent meta-analysis found that only an estimated 59% of participants in North American studies were adherent at a commonly accepted minimal threshold for successful viral suppression [3]. While newer antiretroviral therapy (ART) medications can produce viral suppression at lower levels of adherence, relatively high adherence is still necessary to avoid disease progression and shortened lifespan [4-6]. In addition, low levels of adherence increase the risk of infecting others and contribute to the development of treatment resistant strains of HIV [7;8].

Interventions have been developed to address the significant public health problem presented by poor adherence, with most studies demonstrating some degree of success in the short-term [9]. However, the impact of the interventions is generally not sustained over time [9], and most HIV treatment settings do not have the resources to deliver more intensive interventions. As a result, there has been interest in developing efficacious electronically-delivered interventions. Very little research has focused on establishing the efficacy of mobile health applications for ART adherence. Further, no published studies have examined a single session face-to-face intervention combined with a mobile application and coaching support to reinforce sustained adherence.

Delivered over a smartphone, portable applications would allow for real-time adherence tracking and feedback and ready access to content or services to enhance adherence. The long-term goal of this line of research is to disseminate an efficacious, mobile health ART adherence application that can be integrated readily into clinical care. The objective of this application is to develop a mobile health ART adherence application, to pilot the application, and to conduct a preliminary randomized controlled trial of the application.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed ART, infected with HIV, have a detectable viral load (>20 copies/mL) with the past 6 months, report less than 100% medication adherence, and have a smart phone capable of downloading the mARTAA application.

Exclusion Criteria:

* Physical impairments that prevent completion of the intervention, cognitive impairments that jeopardize informed consent and/or intervention comprehension, active psychosis, and not fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
ART Adherence | 12 Months
  Percentage of ART adherence based on Electronic Pill Box data will be compared between the groups

SECONDARY OUTCOMES:
Self-Reported ART Adherence | 12 Months
  Self-reported ART adherence as measured by the AACTG Medication Adherence Questionnaire will be compared between the groups.
Viral Load | 12 Months
  Viral load will be dichotomized into three levels (20, 48, and 400 copies/ML) and intervention effects will be examined at each of these levels.
Behavioral Skills | 12 Months
  Group differences will be examined in behavioral skills as assessed by the LifeWindows Information-Motivation-Behavioral Skills ART Adherence Questionnaire.
Information | 12 Months
  Group differences will be examined in information as assessed by the LifeWindows Information-Motivation-Behavioral Skills ART Adherence Questionnaire.
Information, Motivation, and Behavioral Skills | 12 Months
  Group differences will be examined in motivation as assessed by the LifeWindows Information-Motivation-Behavioral Skills ART Adherence Questionnaire.
Self-Efficacy | 12 Months
  Group differences will be examined in self-efficacy as assessed by the HIV Treatment Adherence Self-Efficacy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Ramsey, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Ramsey SE, Ames EG, Uber J, Habib S, Clark S, Waldrop D. A Preliminary Test of an mHealth Facilitated Health Coaching Intervention to Improve Medication Adherence among Persons Living with HIV. AIDS Behav. 2021 Nov;25(11):3782-3797. doi: 10.1007/s10461-021-03342-5. Epub 2021 Jun 12. PMID 34117965
- [Derived] Ramsey S, Ames E, Uber J, Habib S, Clark S. A Mobile Health App to Improve HIV Medication Adherence: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2019 Nov 13;8(11):e15356. doi: 10.2196/15356. PMID 31719030